CLINICAL TRIAL: NCT00038805
Title: Allogeneic Stem Cell Transplantation Using Mylotarg (CMA-676) Plus Nonmyeloablative Chemotherapy in Older or Medically Infirm Patients With High-Risk Acute Leukemia (ALL), Chronic Myelogenous Leukemia (CML) or Myelodysplastic Syndrome (MDS)
Brief Title: Nonmyeloablative Preparative Regimen Using Mylotarg for Patients With High Risk Acute Myeloid Leukemia (AML), Acute Lymphocytic Leukemia (ALL), Chronic Myeloid Leukemia (CML) and Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID00-153
Record Dates: First submitted 2002-06-05; First posted 2002-06-07 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Leukemia
Keywords: High Risk Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Chronic Myeloid Leukemia; Myelodysplastic Syndrome; ALL; AML; MDS; CML; CMML; Nonmyeloablative Preparative Regimen; Mylotarg; CMA-676
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mylotarg (Experimental)
  Interventions: Drug: Mylotarg

INTERVENTIONS:
Drug: Mylotarg
  Other Names: CMA-676

SUMMARY:
Primary Objective:

To determine the safety and maximum tolerated dose of CMA-676 as part of an intensive but nonmyeloablative preparative regimen in older or medically infirm patients undergoing mini-allogeneic peripheral blood stem cell transplantation

Secondary Objectives:

1. To evaluate response rates, engraftment kinetics and degree of chimerism achievable with this strategy.
2. To evaluate disease-free and overall survival and relapse rates.
3. To evaluate the need and ability to give multiple cycles of Mylotarg plus FA and mobilized DLI in patients not achieving complete remission.

DETAILED DESCRIPTION:
Mylotarg is a novel immunoconjugate directed against the CD33 antigen found on most leukemia cells. This humanized murine IgG4 monoclonal antibody is tagged with the toxin, calicheamicin. In equal molar concentrations, calicheamicin is about 3200 times more potent than adriamycin. In a Phase I study involving adult patients with relapse AML, Mylotarg has been shown to have significant anti-leukemia activity with little toxicity. The most concerning side effects of Mylotarg were prolonged neutropenia and thrombocytopenia. Phase II studies have also demonstrated good efficacy with little toxicity.

The goal of this proposal is to include Mylotarg in a nonmyeloablative preparative regimen similar to FAI used at MD Anderson Cancer Center. The hypothesis is that Mylotarg will provide potent anti-leukemic effects without adding toxicity to the mini-allogeneic bone marrow transplant regimen. A more potent anti-leukemic response may increase the complete remission rates and induce a state of minimal residual disease (MRD). Therefore, the Graft vs. Leukemia (GVL) effect of allogeneic transplantation will have a better chance for success. In addition, the administration of donor cells after Mylotarg should ameliorate the cytopenias previously associated with Mylotarg. This medication likely will be well-tolerated.

Patients with high-risk hematopoietic malignancies that express CD33 (i.e. AML, ALL, CML and MDS) will be included. We will enroll older patients (>55 years old) or medically infirm patients who are unable to tolerate standard allogeneic bone marrow transplant. Patients will be evaluated at 28 days post-transplant for evidence of response. Those with residual disease may be eligible for additional Mylotarg given together with donor lymphocyte infusions. Additional courses of Mylotarg may improve overall survival in this poor prognosis group.

ELIGIBILITY:
Inclusion Criteria:

* Patients 12-75 years of age
* Patients are eligible if deemed ineligible for conventional high dose chemotherapy programs because of concurrent medical conditions. Patients with refractory AML are eligible provided ejection fraction >= 35%; FEV1, FVC, or DLCO >= 40%; GPT < 3 x normal, direct bilirubin < 2.
* Patients must have recovered from previous Grade III-IV toxicity due to prior antineoplastic therapy (except alopecia).
* Patients with AML with induction failure, relapse or 2nd remission
* Patients with MDS with IPI INT-2 or High-risk disease or CMML.
* Patients with CML in accelerated phase or blast crisis
* Patients with ALL with induction failure, relapse or 2nd remission
* Patients receiving prior BMT are eligible. If myeloablative chemoradiotherapy was used in the prior transplant patients must be >90 days from transplant. If non-myeloablative therapy was used patients must be >30 days post-transplant.
* Leukemia cells must express cell surface CD33 evaluated by flow cytometry in > 20% of leukemia cells.
* Patients must have an HLA identical related donor capable of donating G-CSF stimulated peripheral blood stem cells using apheresis techniques. If patient has a contraindication to PBSC collection bone marrow can be used.
* Patients must have a Zubrod PS <2, Cr <2.0, direct bilirubin <2, and transaminases SGPT <3x normal
* Patients must have an estimated life expectancy > 3 months
* Patient and donor must sign informed consent

Exclusion Criteria:

* no uncontrolled active infection
* no HIV disease
* no pregnancy and no nursing
* no active, uncontrolled CNS leukemia

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2001-05; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of CMA-676 | Continual Reassessment Method (CRM); each cycle

CONTACTS AND LOCATIONS:
Overall Officials: Marcos de Lima, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org